CLINICAL TRIAL: NCT01833910
Title: A Mannequin Study to Assess Various CPR Training Methods Using a Student Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 816764
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest; Heart Disease
Keywords: Cardiopulmonary Resuscitation; Education
MeSH Terms: conditions — Heart Arrest; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Video-only - DVD (Experimental): CPR Training with AHA CPR Anytime DVD presented on a TV with DVD player and no psychomotor skill practice.
  Interventions: Other: AHA CPR Anytime DVD
- Video-only - iPad (Experimental): CPR Training with AHA CPR Anytime DVD presented on a portable video player and no psychomotor skill practice.
  Interventions: Other: AHA CPR Anytime DVD
- Video-only with Household Object (Experimental): CPR Training with AHA CPR Anytime DVD and practice on a household item
  Interventions: Other: AHA CPR Anytime DVD
- Video Self Instruction Kit (Experimental): CPR Training with AHA CPR Anytime Video Self-Instruction kit including manikin
  Interventions: Other: AHA CPR Anytime Video Self-Instruction Kit

INTERVENTIONS:
Other: AHA CPR Anytime Video Self-Instruction Kit — CPR Training utilizing a video self-instruction kit including training video and inflatable manikin.
  Arms: Video Self Instruction Kit
Other: AHA CPR Anytime DVD — A CPR Training Video, originally developed as part of a kit, administered without the accompanying manikin.
  Arms: Video-only - DVD; Video-only - iPad; Video-only with Household Object

SUMMARY:
Prompt delivery of cardiopulmonary resuscitation (CPR) can double a victims chance of survival from cardiac arrest (CA), yet it is provided in less than 1/3 of witnessed events. Studies indicate that video-based education methods can effectively train bystanders in CPR. Using the education and evaluation methods of an existing in-hospital training program, the investigators will assess the CPR skills of students taught with video-only methods, with and without psychomotor skills practice, and compare them to those using a video self-instruction (VSI) kit.

DETAILED DESCRIPTION:
The long term goal of our work is to implement real world CPR training strategies that maximize resuscitation skill retention, and promote willingness to act while addressing major barriers to training including time and cost. To accomplish this, the study team will train student volunteers from the University of Pennsylvania using one of three methods: 1) a video-only method with no psychomotor skill practice, 2) a video-only method with psychomotor skill practice on a household object or 3) a video self-instruction (VSI) kit. Volunteers will be young, healthy students from the University of Pennsylvania with no CPR Training within the last 24 months. The investigators will use the American Heart Association's CPR Anytime Video Self-Instruction Kit which comes equipped with a DVD and inflatable manikin.

For the groups receiving the Video-Only methods, the investigators will remove the inflatable manikin and train the subjects with the DVD. The investigators will randomize the participants to one of the video-only methods or to the VSI kit method of training when they are scheduled for training. Immediately following the training, the investigators will conduct a CPR skills test to measure the effectiveness of the training method. Three (3) to twelve (12) months post-training the investigators will schedule and conduct an in-person interview with subjects. As part of the interview, subjects will be asked to complete a survey measuring their comfort level and willingness to use their CPR skills. Subjects will also be asked to complete another CPR Skills test.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to complete 25-30 minutes of moderate physical activity

Exclusion Criteria:

* CPR Training within the past 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
CPR Compression Quality | 3 months post training
  CPR Compression rate and depth measured on a skill reporting CPR manikin during a simulated cardiac emergency.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Abella, MD, MPhil, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Resusciation Science - Univerity of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Blewer AL, Leary M, Decker CS, Andersen JC, Fredericks AC, Bobrow BJ, Abella BS. Cardiopulmonary resuscitation training of family members before hospital discharge using video self-instruction: a feasibility trial. J Hosp Med. 2011 Sep;6(7):428-32. doi: 10.1002/jhm.847. Epub 2010 Nov 8. PMID 21916007
- [Background] Bobrow BJ, Vadeboncoeur TF, Spaite DW, Potts J, Denninghoff K, Chikani V, Brazil PR, Ramsey B, Abella BS. The effectiveness of ultrabrief and brief educational videos for training lay responders in hands-only cardiopulmonary resuscitation: implications for the future of citizen cardiopulmonary resuscitation training. Circ Cardiovasc Qual Outcomes. 2011 Mar;4(2):220-6. doi: 10.1161/CIRCOUTCOMES.110.959353. Epub 2011 Mar 8. PMID 21386066